CLINICAL TRIAL: NCT05123144
Title: A Stepped Wedge Hybrid Type II Trial of an Online Positive Affect Intervention: Blending Implementation and Effectiveness to Improve HIV Continuum Outcomes in Ryan White Clinics in Chicago
Brief Title: A Hybrid Type II Trial of the Optimizing Resilience and Coping With HIV Through Internet Delivery in Ryan White Clinics in Chicago
Acronym: ORCHID
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Chicago (Other); AIDS Foundation Chicago (Unknown)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: R01MH124632-01 (NIH)
Record Dates: First submitted 2021-06-24; First posted 2021-11-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: People Living With HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Health Screener + ORCHID Intervention (BHS+ORCHID) (Experimental): At the clinic level, sites randomized to implement BHS+ORCHID will receive training, materials, and other support to administer behavioral health screening and refer their clients with elevated depression symptoms to ORCHID.
  At the individual level, those clients who are eligible and choose to enroll in ORCHID will receive self-guided training on 8 positive affect skills through weekly online sessions and daily practice exercises.
  Interventions: Behavioral: BHS+ORCHID
- Standard of Care (No Intervention): usual care

INTERVENTIONS:
Behavioral: BHS+ORCHID — At the clinic level, sites randomized to implement BHS+ORCHID will receive training, materials, and other support to administer behavioral health screening and refer their clients with elevated depression symptoms to ORCHID.
  At the individual level, those clients who are eligible and choose to enroll in ORCHID will receive self-guided training on 8 positive affect skills through weekly online sessions and daily practice exercises.
  Arms: Behavioral Health Screener + ORCHID Intervention (BHS+ORCHID)

SUMMARY:
Among people living with HIV (PLWH), positive affect is uniquely associated with lower levels of depression, slower disease progression, better adherence to medication, and higher likelihood of achieving suppressed viral load, independent of negative affect. In two randomized controlled trials with PLWH (R01 MH084723; R01 DA033854), the investigators have shown significant beneficial effects of an intervention that aims to increase positive affect on viral suppression and psychological well being. The investigators also have demonstrated feasibility, acceptability, and early efficacy of a self-guided, online-delivered, positive affect skills intervention for PLWH (R34 MH101265). Now, in collaboration with the AIDS Foundation of Chicago (AFC), the investigators propose to conduct a Hybrid Type II effectiveness-implementations study of a stepped wedge cluster randomized trial (SW-CRT) of mental health screening and referral to ORCHID (Optimizing Resilience and Coping with HIV through Internet Delivery). The proposed study was initiated by AFC, which developed the mental health screening and selected the SW-CRT design as an ethical way to study implementation while ensuring that all clients with elevated depression receive the intervention. Mental health screening + ORCHID will be implemented through all medical case managers (MCMs) at 17 Ryan White-funded clinics in Chicago. The investigators will use the RE-AIM framework to structure the effectiveness and implementation outcomes and the Consolidated Framework for Implementation Research (CFIR) to understand the implementation outcomes at the patient and clinic levels. The specific aims are to: (1) Operationalize an implementation facilitation strategy to link mental health screening with referral to ORCHID through MCMs at Ryan White-funded clinics in Chicago; (2) Determine the effectiveness of screening + ORCHID for improving depression, retention in care, and viral suppression, among 300 PLWH receiving care at 17 Ryan White clinical sites, using a stepped wedge cluster randomized design. Depression is the primary outcome and retention in care and viral suppression at both the individual and clinic level are the secondary outcomes; and (3) Evaluate the implementation of screening + ORCHID and iteratively refine the strategy for subsequent steps. The proposed research holds significant promise for advancing current knowledge on how best to integrate and respond to mental health screening in Ryan White clinics. Data from the hybrid trial will result in a sustainable, scalable program that can be disseminated in Ryan White clinics nationwide, thus holding significant promise for advancing Chicago toward goals in the National Ending the HIV Epidemic Plan.

DETAILED DESCRIPTION:
Current HIV prevention strategies for PLWH emphasize engagement across the HIV Continuum of Care: linkage to and retention in care, adherence to antiretroviral therapy, and maintenance of suppressed viral load. The National HIV/AIDS Strategy goals for engagement in each phase of the continuum include: 85% of those diagnosed with HIV linked to care within 1 month, 90% of those living with HIV retained in care, and 80% achieving suppressed viral load.23 As with many other cities, Chicago falls far below these targets: in 2018, only 41.1% of PLWH were retained in care, as measured by having at least 2 visits during which CD4 or viral load count were obtained 3 months apart, and 52% were virally suppressed (i.e., <200 copies/mL at their last viral load test).

Depression, highly prevalent in PLWH, predicts HIV progression and is associated with lack of engagement in Continuum of Care. Screening for depression is a first step to addressing the significant barrier to engaging in care and improving the health and well-being of PLWH. However, even if clients are routinely screened, there are few models of effective, sustainable, and cost-effective mental health care that are easily integrated into clinic workflow. In many places, there is a dearth of mental health providers and services able to address the needs of PLWH and depression. The investigators propose to address this gap with ORCHID (Optimizing Resilience and Coping with HIV through Internet Delivery), a self-guided online-delivered intervention that specifically targets positive affect. The theory and empirically-based program includes eight skills (noticing and capitalizing on positive events, gratitude, mindfulness, positive reappraisal, personal strengths, attainable goals, and self-compassion), delivered in a self-guided online format. Across delivery modes and type of participant stress, the intervention has shown good feasibility, acceptability, and efficacy.

The intervention is based on revised Stress and Coping Theory and the Broaden-and-Build Theory of positive emotion. The preliminary data for the proposed study consists of 1) two randomized trials of an in-person positive affect intervention for PLWH who are newly diagnosed (n=159) or are sexual minority men who use methamphetamines (n=110); 2) an online adaptation of the positive affect intervention for people with elevated depression demonstrates feasibility, acceptability and efficacy (n=539); and 3) a pilot RCT of the online version of this intervention conducted with 21 PLWH.

The goal of the proposed study is to examine whether those who complete ORCHID, as implemented through Ryan White clinics, will experience improvements to depression and engagement in care. At the clinic level, we will examine whether clinics that are implementing the screening and referral to ORCHID have overall lower depression and higher engagement in care, compared to those clinics not yet implementing the screening and ORCHID referral. If effective, the ORCHID program can be disseminated to other geographical locations facing a high burden of HIV.

ELIGIBILITY:
Inclusion Criteria:

Clinic-Level:

* Ryan White clinic in the Chicagoland area
* On-site medical services

Individual-Level:

* Age 18 and over
* Speaks and reads English
* Receives medical case management through one of the eligible Ryan White clinics
* Referral from medical case manager (on basis of screening positive for elevated depression through a clinic-based screener; PHQ-9 score > 5)
* Daily access to a device connected to the internet
* Willingness to provide access to health and medical care from the Chicago Department of Health, primary care provider, and/or from the AIDS Foundation Chicago, confirmed by signature on two Release of Information forms.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | 12 months
  Primary outcome is change on depression (PROMIS-depression) from baseline to the 3 follow up points out to 12 months post intervention

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AIDS Foundation of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Based on the updated NIH Policy as of January 2018, we aim to make the data available as early as 12 months after primary data collection has been completed depending on the study timeline and research team's progress on data collection, rigorous data analysis, consultation with field experts/collaborators, manuscript writing, and timing of publication.

REFERENCES:
- [Derived] Garner BR, Bouris A, Charlebois ED, Li DH, Dakin A, Moskowitz J, Benbow N, Christopoulos K, Hickey MD, Imbert E. The Strategies Timeline and Activities Reporting Tables: Improving HIV Care by Improving the Reporting of Implementation Strategies. J Acquir Immune Defic Syndr. 2025 Apr 15;98(5S):e205-e215. doi: 10.1097/QAI.0000000000003613. PMID 40163072
- [Derived] Xavier Hall CD, Ethier K, Cummings P, Freeman A, Bovbjerg K, Bannon J, Dakin A, Abujado F, Bouacha N, Derricotte D, Patterson L, Hirschhorn LR, Bouris A, Moskowitz JT. A hybrid type II effectiveness-implementation trial of a positive emotion regulation intervention among people living with HIV engaged in Ryan White Medical Case Management: protocol and design for the ORCHID study. Trials. 2024 Sep 27;25(1):631. doi: 10.1186/s13063-024-08475-1. PMID 39334472